CLINICAL TRIAL: NCT07083882
Title: Faecal Autologous Capsule Transplantation for Type 1 Diabetes Mellitus
Acronym: FACT-T1D
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Diabeter Centrum Amsterdam (Unknown)
Responsible Party: Principal Investigator, Nordin Hanssen, Associate Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: METC2025.0067
Record Dates: First submitted 2025-07-11; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes Mellitis; Type 1 Diabetes (T1D); Fecal Microbiota Therapy (FMT)
Keywords: microbiome; type 1 diabetes; microbiota transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: placebo matching capsule without microbial content
- Encapsulated autologous fecal microbiota transplantation (Experimental)
  Interventions: Biological: freezedried autologous encapsulated fecal microbiota transplantation

INTERVENTIONS:
Biological: freezedried autologous encapsulated fecal microbiota transplantation — The freezedried autologous encapsulated microbiota transplantation increases the exposure of the small intestine to the microbiota residing in the colon. Prior evidence was found that this has strong immunomodulatory effects leading to potential preservation of beta cell function in type 1 diabetes.
  Arms: Encapsulated autologous fecal microbiota transplantation
Other: placebo matching capsule without microbial content — this is the matching placebo capsule that looks from the outside identical to the actual treatment but does not contain the fecal microbiota.
  Arms: Placebo

SUMMARY:
SUMMARY

Rationale:

The(small) intestinal microbiota composition has been implicated to play an important role in (human) metabolism, as well as autoimmune diseases such as type 1 diabetes mellitus. Faecal microbiota transplantation (FMT) has been shown to significantly alter the microbiota composition, without any serious side-effects. It was recently demonstrated that multiple infusions of own faeces(autologous) preserved residual beta cell function up to one year after start of the FMT. In a proof-of-principle study it was found that encapsulated autologous FMT provides a safe and feasible option for prolonged treatment on a daily basis, which might stabilize the beta-cell destruction. These exciting findings are potentially transformative for clinical practice and deserve replication in a larger placebo-controlled trial.

Objective: confirm the efficacy and feasibility of daily ingested encapsulated freeze-dried autologous (own)faecal matter on the preservation of residual beta cell function as assessed by C-peptide release upon amixed meal test (MMT) in recently diagnosed type 1 diabetes mellitus (T1D).

Study design: double-blind placebo-controlled study Study population: n=110, recently diagnosed (<100 days of diagnosis) patients with T1D, aged 18-45 years, BMI 18-30 kg/m2, male/female.

Intervention: After inclusion and randomisation individuals will receive for 6 months either placebo or freeze-dried autologous encapsulated FMT in a 1:2 ratio. Subsequently, participants with be followed for 6 months whether beta cell preservation was durable after cessation of treatment.

Main study parameters/endpoints: The primary endpoint is long-term preservation of beta cell insulin secretion capacity as assessed by stimulated C-peptide AUC0-120minresponse upon MMT (at0, 6 and 12months).The secondary endpoint pertains to changes in post-meal urinary C-peptide levels, plasma biochemistry (HbA1c levels),glucose time-in-range and subsequentexogenous insulin dose use at 0, 6 and 12months.

Nature and extent of the burden and risks associated with participation,benefit and group relatedness: This study is considered a low-risk study, 3MMTs will be performed, for which 70 ml of blood samples will be drawn each visit. As of today, no severe adverse events as result of FMT have been reported in this centre and in the ENCAPSULATE trial investigating the feasibility and safety of this approach participants only reported some minor and transient constipation. In addition, the use of autologous faeces comes with a lower(absent)risk for transmitting any unknown pathogens compared to an allogenic FMT. As there currently is no widely applied therapy to preserve beta cell function in type 1 diabetes, encapsulated autologous FMT can have a potential benefit for the participants.

DETAILED DESCRIPTION:
OBJECTIVES This study is designed to confirm whether a microbial intervention based on capsules containing autologous (own) lyophilized faecal microbiota, LFMCs, taken daily for 6 months has beneficial effects on residual beta cell function (C-peptide secretion uponMMT) in recently diagnosed type 1 diabetes mellitus compared to placebo. A parallel objective is to assess the impact on glycaemic control.

To investigate the effect of daily oral intake of autologous LFMCs on:

I Preservation of residual beta cell insulin secretion capacity: assessed by maximal C-peptiderelease(residual beta cell function)upon an MMT, AUC0-120min at 0,6 and 12 months. As an additional marker of residual beta cell function, at home post-meal urinary C-peptide levels will be used.

II Glycaemic control: changes in plasma biochemistry (glucose, HbA1c), glucose time in range (FreestyleLibre), urine (microalbuminuria) and subsequent exogenous insulin dose use at 0,6 and 12months.

III Questionnaires and dietary intake: validated questionnaires for abdominal complaints, diabetic complications and hypoglycaemia frequency at 0,6 and 12 months. Dietary intake will be registered via online dietary lists at 0,6 and 12months.

STUDY DESIGN This is a placebo controlled, double blind, single-centre study. After the randomisation, in a 1:2 (placebo:LFMC) ratio using a validated variable block randomization model in Castor, stratified for sex with block sizes 4,6 and 8, participants will ingest the autologous LFMCs or placebo daily for 6months, which will be followed by a follow-up period of 6months. In total, participants will be followed for12months after inclusion.

Study visits Subjects will in principle visit 3 times in total for this study, with 1 prior screening visit that essentially encompasses participation in the MARVEL cohort (NL85375.018.23, measuring residual beta cell function and questionnaires) and one visit to pick up the second batch of capsules. Each visit will take 180 minutes (maximum of 12 hours over 12 months).

Screening Blood will be drawn for basic biochemistry and patients will hand in the food diaries, questionnaires. In addition, height, weight, blood pressure will be measured and BMI will be calculated. As the faeces is needed to produce the autologous LFMCs, participants are instructed to collect at least 300 grams of fresh faeces. If the fresh faeces is insufficient (<300g), participants are asked to collect more fresh faeces and bring thisto the AMC at a later date (but before the baseline visit).

Optional: additional fecal collections. It may be the case that individuals produce insufficient feces at once, in that case participants are asked to bring in addition samples until 300g is reached.

Visit1: baseline visit (0 months) At baseline a MMT will be performed, blood will be drawn for basic biochemistry and patients will hand in the food diaries, questionnaires and their fecal and 2h post-meal urine sample. Thereafter, the participant will start with the LFMCs for 6months. The first capsule is ingested with the investigator present to ensure the participant tolerates the capsules well and has an appropriate intake technique.

Visit 2 (3months): by phone to evaluate compliance and potential side-effects.

Visit3: follow-up visit (6months) During this visit the MMT will be repeated, blood will be drawn for basic biochemistry and patients will hand in the food diaries and questionnaires and their 2h post-meal urine sample. In addition, height, weight, blood pressure are measured again. Participants stop with the LFMCs and return any remaining capsules to the investigator.

Visit4: follow-up visit (12months) During this last visit, the MMT will berepeated, blood will be drawn for basic biochemistry and patients will hand in the food diaries, questionnaires and their 2h post-meal urine sample. In addition, height, weight, blood pressure are measured again.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female recently diagnosed (<100 days) with type 1 diabetes mellitus.
2. Age:18-45 years
3. BMI: 18-30 kg/m2
4. Remaining residual beta cell function: detectable plasma C-peptide or urinary C-peptide at inclusion of the study.

Exclusion Criteria:

1. Major systemic illness
2. (Expected) prolonged comprised immunity (e.g. due to recent cytotoxic chemotherapy or human immunodeficiency virus(HIV) infection with a CD4 count < 240/mm3).
3. History of a severe disease of the digestive tract, such as celiac disease, chronic diarrhoea (≥3 stools/day for >4 weeks), chronic obstipation (<2 defecations/week for >3 months) or Inflammatory Bowel Disease (IBD).
4. Illicit drug use (e.g. MDMA/amphetamine/cocaine/heroin/GHB) in the past three months or use during the study period.
5. Use of >21 units of alcohol per week on average in the past three months.
6. Pregnancy or breast feeding.
7. Inability to provide informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Preservation of residual beta cell insulin secretion capacity | At baseline, at 6 months upon completion of treatment and at 12 months after intiation of treatment
  measured by plasma C-peptide in mixed meal and 2hour post meal urine sample

SECONDARY OUTCOMES:
Hba1c | At baseline, at 6 months upon completion of treatment and at 12 months after intiation of treatment
  expressed as mmol-mol
Continuous glucose monitoring | At baseline, at 6 months upon completion of treatment and at 12 months after intiation of treatment
  Time in range expressed as % and time below range expressed as %
albuminuria | At baseline, at 6 months upon completion of treatment and at 12 months after intiation of treatment
  expressed as ratio urinary albumin an kreatinin, as mg-mol
exogenous insulin dose | At baseline, at 6 months upon completion of treatment and at 12 months after intiation of treatment
  expressed as units used per 24 hours

OTHER OUTCOMES:
GI-Symptoms Rating Scale (GSRS) | At baseline, at 6 months upon completion of treatment and at 12 months after intiation of treatment
  The GSRS is a commonly used questionnaire about the presence of gastrointestinal symptoms and consists of fifteen questions that correspond to five different abdominal syndromes scored 1 (no symptoms) to 7 (most severe complaints). If all syndromes are below 3 no symptoms is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Diabeter Centrum Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No